CLINICAL TRIAL: NCT01917474
Title: Effects of Changes in Dietary Intake and Headache's Attacks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ferrara Liberato Aldo, Associate Professor of Medicine, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Headache
Keywords: low-lipid diet; normal lipid intake; saturated fats reduction; headache attacks
MeSH Terms: conditions — Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Low-lipid diet (Experimental): Lifestyle counseling At the end of this run-in period all patients will be randomly attributed to one of the following two dietary regimens. Those in the experimental groupwill be given a low lipid diet with a lipid content < 20% of the total daily energy intake with the following composition:
  Proteins (g) 77 (15% total energy intake) Lipids (g) 48 (22% total energy intake) Saturated (g) 9 (4% total energy intake) Monounsaturated (g) 31 (14% total energy intake) Polyunsaturated (g) 8 (4% total energy intake) Carbohydrates (g) 330 (63% total energy intake) Cholesterol (mg) 117 Fibres (g) 32 Total Energy (kcal) 1977
  Interventions: Dietary Supplement: low lipid diet; Dietary Supplement: normal lipid diet
- normal lipid diet (Active Comparator): Patients in the active comparator will be given a diet with normal lipid intake and the following composition:
  Proteins (g) 75 (15% total energy intake) Lipids (g) 67 (29% total energy intake) Saturated (g) 14 (6% total energy intake) Monounsaturated (g) 43 (19% total energy intake) Polyunsaturated (g) 10 (4% total energy intake) Carbohydrates (g) 307 (56% total energy intake) Cholesterol (mg) 128 Fibres (g) 32 Total Energy (kcal) 2048 lipid intake between 25-30% of the total daily energy intake.
  Interventions: Dietary Supplement: low lipid diet; Dietary Supplement: normal lipid diet

INTERVENTIONS:
Dietary Supplement: low lipid diet — Patients will receive a diet of about 2000 kcal daily with no more than 20 % of the total energy coming from lipids, mainly from the monounsaturated olive oil
Dietary Supplement: normal lipid diet — Patients will receive a diet of about 2000 kcal daily with 28 % of the total energy coming from lipids, mainly from the monounsaturated olive oil

SUMMARY:
Headache is a frequently disabling disorder, which occurs in about 30% of the adult population, particularly in overweight/obese women. Aim of the study is to modify the nutritional habits of the patients and to evaluate the effects of a low lipid intake vs. a normal lipid diet on the incidence and severity of migraine crises. Moreover vascular reactivity will be evaluated in a randomly selected subgroup of patients. This randomized, cross-over intervention trial will be performed in about 150 patients, affected by migraine. Adherence to the diet, particularly regarding energy intake, percent of energy from lipids, carbohydrates and proteins will be carefully assessed at baseline and during the 2 intervention periods

DETAILED DESCRIPTION:
Headache is a common disease in general population, which affects adult women more frequently than men. Among different factors which might be involved in the pathophysiology of the disease, eating or drinking a particular food or drink have been shown to act as a trigger of acute attacks. In particular foods such as aged cheese or red wine may trigger acute migraine attacks and dietary habits such as excessive caffeine intake may increase headache frequency.

Moreover a close relationship has been detected between overweight/obesity and migraine severity even if other authors showed that obesity at baseline does not seem to be related to follow-up refractoriness to preventive treatment.

At the first visit, patients will undergo a complete clinical examination and body weight (BW), height (HT), blood pressure (SBP/DBP) and heart rate (HR) will be also measured. Body mass index (BMI) will be calculated as BW/HT2 and expressed in kg/m2. We consider overweight patients with BMI> 25 and < 30 whilst frankly obese are those with BMI > 30. Patients will be followed-up for two months when treatment for the prevention of headache (usually the calcium entry blocker flunarizine 5 mg/day) will be added to the habitual dietary regimen. At the end of this run-in period all patients will be randomly attributed to one of the following two dietary regimens: a low lipid diet with a lipid content < 20% of the total daily energy intake and a normal lipid diet with a lipid intake between 25-30% of the total daily energy intake. In both diet lipid intake is mostly represented by monounsaturated fatty acids (14% in the low lipid and 19% in the normal lipid diet) with a low intake of saturated fats (< 8%of the total calories, which is the percentage usually recommend in our diets). Patients will be followed-up for 2 months at the end of which they will be switched to the alternative dietary regimen.

At baseline and during the observation period patients will be seen at the Headache Outpatient Clinic of our department at one month intervals. At each visit they will be given a form to be filled at home, summarizing the number of the monthly headache attacks, the severity of each one graded from 0.1 to 3 from mild to severe pain, and how many times they assumed pills for the therapy of the attacks during the last month. Headache attacks with severe pain will be considered those receiving a score > 2.5. Moreover, at each visit patients will fill-up a food questionnaire, validated in comparison to the 7-day food record (12), with the help of a well trained dietician. Data are expressed as daily percent caloric intake from each macronutrient and as the weekly number of a medium size serving.

Main drugs suggested for the pain relief at each attack are the selective serotonin receptor agonists (triptans), which are abortive migraine medications, and the non steroidal anti-inflammatory agents.

In a randomly selected subgroup of patients we will evaluate at baseline and after diet:

1. Vascular dysfunction by echography at the brachial artery level after ischaemia (Flow mediated dilatation) and after nitroglycerin 0.3 mg;
2. Intimal-media thickness at carotid artery level will be evaluated by b-mode echography;
3. central pressure and pulse wave velocity by tonometry applanation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary headache on free diet

Exclusion Criteria:

* Patients with laboratory or TC findings of secondary headache

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
To verify the possibility that low-lipid diet might reduce of the half the number and intensity of headache attacks.It will be considered efficacy if will be a reduction of 50% of headheach crisis after two months of dietetic low lipid treatment | after 2-months of dietary treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liberato A ferrara, MD, Principal Investigator — Dept. of Medicine and Surgery; Federico 2nd University of Naples
Locations (2):
- Italy (2):
  - Federico 2nd University of Naples, Naples
  - Headache Outpatient Clinic Dept. of Clinica Medica; Federico 2nd University of Naples, Naples

REFERENCES:
- [Derived] Ferrara LA, Pacioni D, Di Fronzo V, Russo BF, Speranza E, Carlino V, Gargiulo F, Ferrara F. Low-lipid diet reduces frequency and severity of acute migraine attacks. Nutr Metab Cardiovasc Dis. 2015 Apr;25(4):370-5. doi: 10.1016/j.numecd.2014.12.006. Epub 2014 Dec 27. PMID 25698152